CLINICAL TRIAL: NCT05693883
Title: The Effects of Pilates Training on Symptoms in Patients With Allergic Rhinitis
Brief Title: Pilates Training in Patients With Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Wannaporn Tongtako, Ph.D., Principal investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ex Physio SPSC 4
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis; Pilates; Cytokine; Pulmonary function; Rhinitis symptoms
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates training (Experimental): The participant completed receiving pilates training program three time a week for ten week-long (60 minutes/time)
  Interventions: Other: Pilates training
- Control group (No Intervention)

INTERVENTIONS:
Other: Pilates training — Subject participating in 60-min sessions for 10 weeks and Each session consisted of a 10-min warm up (Breathing, Imprint & release, Hip release, Spine rotation, Hip rolls, Scapula isolation, Arm circle, Elevation & depression scapulae, Head nod, Cat stretch), Pilates program 40-min (Toe tap, Ad prep, Breast stroke preps, Heel squeeze prone, Side leg lift, Single leg extension, One leg circle, Shoulder bridge prep, Four point, kneeling, Spine twist, Hundred prep, Roll up prep, shoulder bridge prep2, Breast stroke, Swimming, Half roll back) and 10-min cool down (Spine stretch forward, Shell stretch, Side bending, Cat stretch, Roll down)
  Arms: Pilates training

SUMMARY:
The purpose of this study was to determine the effects of pilates training on symptoms in patients with allergic rhinitis.

DETAILED DESCRIPTION:
Twenty allergic rhinitis patients aged 18 - 35 years were randomized into 2 groups: control group (CON; n=9) and pilates training group (PTG; n=11). Participants in CON group do their daily routine without receiving any training program, while those in PTG group completed receiving pilates training program three time a week for ten week-long (60 minutes/time). The physiological data, rhinitis symptoms, cytokines, pulmonary function, respiratory muscle strength were analyzed during the pre-test and post-tests. The dependent variables between pre-test and post-tests were analyzed by paired t-test. The rhinitis symptoms and cytokines variables between pre-test and post-test were analyzed by repeated measures ANOVA. In addition, an independent t-test was used to compare the variables between groups. Statistical significance was defined as p < .05.

ELIGIBILITY:
Inclusion Criteria:

* the persistent allergic rhinitis who had rhinitis symptoms more than 4 days a week and positive skin prick test to house dust mite were recruited
* stopped taking all medicine before the study sus as antihistamine for 3 days, oral steroid and nasal steroid for at least 2 weeks and leukotriene receptor antagonist for at least a week prior to the study
* had no exercise program, non-smoking and without any food supplementation for at least 6 months prior to the start of the study

Exclusion Criteria:

* had complications with allergic rhinitis, sinusitis, ear tube malfunctions, asthma, lung cancer, emphysema, lower back pain, tendinitis and arthritis

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Rhinitis symptom scores | Change from Baseline Rhinitis symptom scores at 10 weeks.
  Nasal symptoms were assessed using Total Nasal Symptom Score (TNSS) questionnaire. The subjects were asked to score symptoms of persistent allergic rhinitis before and after yoga training protocol. The total nasal symptom scores were computed as the sum of four individual nasal symptom scores; nasal congestion, itching, sneezing, and rhinorrhea. The scores ranged from 0 to 3 scale (0=none, 1=mild, 2=moderate, 3= severe)
Cytokine in nasal secretion | Change from Baseline cytokines scores at 10 weeks.
  Nasal secretions collection was performed bilaterally with filter paper strips (7x30 mm Whatman No.42, Whatman, Clifton, NJ). Three filter paper strips were sequentially placed on each anterior portion of the inferior turbinate for 10 min. This filter paper strips were collected into appropriate tubes and centrifuged at 3,000 rpm for 5 min at 4 °C and immediately frozen at -70 °C until later analysis.The levels of cytokines were determined by using Sandwich ELISA technique

SECONDARY OUTCOMES:
Respiratory muscle strength change | Change from Baseline respiratory muscle strength at 10 weeks.
  Respiratory muscle strength was assessed by measuring Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) in cmH2O. The participants were in a sitting position using a portable handheld mouth pressure meter (i.e., MicroRPM) with a nose clip. For the MIP measurement, the participants were asked to exhale until they felt no air remaining in their lungs (starting with the functional residual capacity [FRC] point), then held the device on their mouth and inhaled forcefully for 1-2 seconds. For the MEP measurement, the participants were asked to inhale until their lungs were completely filled with air (starting with the total lung capacity [TLC] point), then they kept the device on their mouth and exhaled forcefully for 1-2 seconds
Pulmonary Functions | Change from Baseline Pulmonary Functions at 10 weeks.
  The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration.

CONTACTS AND LOCATIONS:
Overall Officials: Wannaporn Tongtako, Ph.D., Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Sports Science, Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franco CB, Ribeiro AF, Morcillo AM, Zambon MP, Almeida MB, Rozov T. Air stacking: effects of Pilates mat exercises on muscle strength and on pulmonary function in patients with cystic fibrosis. J Bras Pneumol. 2014 Oct;40(5):521-7. doi: 10.1590/s1806-37132014000500008. PMID 25410840
- [Result] Barbosa AW, Guedes CA, Bonifacio DN, de Fatima Silva A, Martins FL, Almeida Barbosa MC. The Pilates breathing technique increases the electromyographic amplitude level of the deep abdominal muscles in untrained people. J Bodyw Mov Ther. 2015 Jan;19(1):57-61. doi: 10.1016/j.jbmt.2014.05.011. Epub 2014 Jun 5. PMID 25603743
- [Result] Brozek JL, Bousquet J, Agache I, Agarwal A, Bachert C, Bosnic-Anticevich S, Brignardello-Petersen R, Canonica GW, Casale T, Chavannes NH, Correia de Sousa J, Cruz AA, Cuello-Garcia CA, Demoly P, Dykewicz M, Etxeandia-Ikobaltzeta I, Florez ID, Fokkens W, Fonseca J, Hellings PW, Klimek L, Kowalski S, Kuna P, Laisaar KT, Larenas-Linnemann DE, Lodrup Carlsen KC, Manning PJ, Meltzer E, Mullol J, Muraro A, O'Hehir R, Ohta K, Panzner P, Papadopoulos N, Park HS, Passalacqua G, Pawankar R, Price D, Riva JJ, Roldan Y, Ryan D, Sadeghirad B, Samolinski B, Schmid-Grendelmeier P, Sheikh A, Togias A, Valero A, Valiulis A, Valovirta E, Ventresca M, Wallace D, Waserman S, Wickman M, Wiercioch W, Yepes-Nunez JJ, Zhang L, Zhang Y, Zidarn M, Zuberbier T, Schunemann HJ. Allergic Rhinitis and its Impact on Asthma (ARIA) guidelines-2016 revision. J Allergy Clin Immunol. 2017 Oct;140(4):950-958. doi: 10.1016/j.jaci.2017.03.050. Epub 2017 Jun 8. PMID 28602936
- [Result] Chanta A, Klaewsongkram J, Mickleborough TD, Tongtako W. Effect of Hatha yoga training on rhinitis symptoms and cytokines in allergic rhinitis patients. Asian Pac J Allergy Immunol. 2022 Jun;40(2):126-133. doi: 10.12932/AP-260419-0547. PMID 31421665